CLINICAL TRIAL: NCT01585038
Title: A Randomized Controlled Trial Comparing Efavirenz With Rilpivirine on Changes in Endothelial Function, Inflammatory Markers, and Oxidative Stress in HIV-uninfected Healthy Volunteers
Brief Title: Efavirenz Versus Rilpivirine on Vascular Function, Inflammation, and Oxidative Stress
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Janssen Services, LLC (Industry)
Responsible Party: Principal Investigator, Samir K Gupta, MD, MS, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMC278HIV4002
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Results first posted 2015-07-02 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-07

CONDITIONS: Cardiovascular Disease
Keywords: endothelium; inflammation; oxidative stress; HIV-1
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation | interventions — efavirenz; Rilpivirine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Efavirenz (Active Comparator): Efavirenz 600mg given nightly without food for 30 days
  Interventions: Drug: Efavirenz
- Rilpivirine (Active Comparator): Rilpivirine 25mg given daily with meals for 30 days
  Interventions: Drug: Rilpivirine

INTERVENTIONS:
Drug: Efavirenz — 600mg orally every evening
  Other Names: Sustiva, Stocrin
  Arms: Efavirenz
Drug: Rilpivirine — 25mg orally once daily
  Other Names: Edurant
  Arms: Rilpivirine

SUMMARY:
The purpose of this study is to compare the cardiovascular profiles of efavirenz and rilpivirine, which are two drugs used to treat HIV infection.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label, single-center study comparing the effects of efavirenz (EFV) versus rilpivirine (RPV) on endothelial function in a total of 40 HIV-uninfected healthy volunteers (20 in each arm) at the Indiana University Medical Center. Enrolled subjects will have their brachial artery flow-mediated dilation (FMD), a measure of endothelial function, and other cardiovascular, inflammatory, and oxidative stress parameters measured at baseline and again after 4 weeks of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Negative ELISA for HIV-1 or HIV-2 at screening
3. Negative hepatitis B surface antigen at screening
4. Negative hepatitis C antibody at screening
5. For women of reproductive potential, a negative urine pregnancy test at screening and willingness to use two forms of birth control during the course of the study
6. For men who are capable of impregnating a female sexual partner, a willingness to use condoms with spermicidal gel for all sexual contacts during the course of the study
7. No documented history of or receipt of medications being used to treat any psychiatric disorder, including (but not limited to) depression, dysthymia, mania, bipolar disease, schizophrenia, or previous suicidal ideation/attempts
8. No anticipated changes or additions to other medical therapies during the course of the study
9. No documented history of seizure disorder

Exclusion Criteria:

1. Inability to provide written, informed consent
2. Known allergy/intolerance to rilpivirine, efavirenz, or nitroglycerin
3. Absolute neutrophil count < 750cell/mL at screening
4. Hemoglobin < 11g/dL at screening
5. Platelet count < 100,000/mL at screening
6. Estimated creatinine clearance (per Cockcroft-Gault equation) < 55 mL/min at screening
7. Liver transaminases (AST or ALT) > 100 IU/mL or total bilirubin > 1.5mg/dL at screening
8. Serum glucose > 200mg/dL at screening
9. Serum total cholesterol > 190mg/dL at screening
10. Breastfeeding at screening or during the course of the study
11. Hypotension, defined as SBP < 90mmHg at time of each main study visit before brachial artery ultrasound measurements
12. Hypertension, defined as SBP > 160mmHg at time of screening
13. Receipt of investigational agents within 30 days of each screening visit or anticipated use during the trial
14. Receipt of cytotoxic chemotherapy within 30 days of each screening visit or anticipated use during the trial
15. Receipt of systemic glucocorticoids (> 10mg/day of prednisone or the equivalent), inhaled/nasal/topical fluticasone, or anabolic steroids within 30 days of each screening visit or anticipated use during the trial
16. Use of sildenafil (Viagra or Silagra), vardenafil (Levitra), or tadalafil (Cialis), within 72 hours (before or after) of brachial artery reactivity testing
17. Indwelling vascular catheters within any upper body vessel at time of brachial artery reactivity testing
18. Active drug or alcohol use or dependence that, in the opinion of the investigator or study personnel, would interfere with adherence to study requirements
19. Acute therapy for serious infection or other serious medical illnesses (in the judgment of the site investigator) requiring systemic treatment and/or hospitalization within 14 days prior to each screening and study visit
20. History of migraine headaches
21. History of Raynaud's phenomenon
22. History of cardiac arrythmias
23. History of hypothyroidism or hyperthyroidism that is untreated (defined as a TSH outside the normal range on most recent testing during normal clinical care)
24. History of carotid bruits
25. History of any tobacco use (cigarette smoking, cigar smoking, chewing tobacco) or nicotine replacement treatments (patch, gum) within 45 days of screening
26. Drugs/therapies with significant CYP 450 induction or inhibition potential at screening
27. Use of antacids, H2-blockers, or proton pump inhibitors within 30 days of screening or anticipated use of these drugs during the trial
28. Any history of injection or illicit drug use
29. Presence of fever, defined as an oral or tympanic temperature > 100.3F, at either the Entry or Closeout Visits
30. On the PHQ-9 depression questionnaire at screening, a total score of more than 9 or any score over 0 on question 9.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir K Gupta, MD, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana Clinical and Translational Sciences Institute, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Gupta SK, Slaven JE, Kamendulis LM, Liu Z. A randomized, controlled trial of the effect of rilpivirine versus efavirenz on cardiovascular risk in healthy volunteers. J Antimicrob Chemother. 2015 Oct;70(10):2889-93. doi: 10.1093/jac/dkv195. Epub 2015 Jul 13. PMID 26169561

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Efavirenz | Rilpivirine
Started | 20 | 20
Completed | 18 | 18
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Efavirenz | Rilpivirine | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Full Range); unit: years] | 30.4 [20.3 to 54.5] | 34.5 [20.4 to 66.3] | 31.54 [20.33 to 66.33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 5 | 10 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 17 | 19 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Flow-mediated Dilation of the Brachial Artery
Description: This is a measure of in vivo endothelial function
Time Frame: Change from baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: absolute percentage change
Arm/Group | Efavirenz | Rilpivirine
Number analyzed (Participants) | 18 | 18
absolute percentage change | 0.089 (3.65) | 0.63 (2.42)
Statistical Analysis 1: Comparison: Efavirenz vs Rilpivirine; Test type: Superiority or Other; p = 0.30, t-test, 1 sided; Mean Difference (Net) = 0.54, 95% CI 2-sided [-1.56 to 2.64]

2. Secondary Outcome: Inflammatory Markers
Description: Change in high sensitivity C-reactive protein levels
Time Frame: Change from baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Efavirenz | Rilpivirine
Number analyzed (Participants) | 18 | 18
mg/L | 0.80 (2.47) | -0.41 (6.01)
Statistical Analysis 1: Comparison: Efavirenz vs Rilpivirine; Test type: Superiority or Other; p = 0.35, t-test, 2 sided; Mean Difference (Net) = -1.21, 95% CI 2-sided [-4.71 to 2.30]

3. Secondary Outcome: Endothelial Activation Markers
Description: Change in soluble vascular cell adhesion molecule-1 levels
Time Frame: Change from baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Efavirenz | Rilpivirine
Number analyzed (Participants) | 18 | 18
pg/mL | -27.62 (125.20) | -20.92 (68.95)
Statistical Analysis 1: Comparison: Efavirenz vs Rilpivirine; Test type: Superiority or Other; p = 0.41, t-test, 2 sided; Mean Difference (Net) = 6.70, 95% CI 2-sided [-62.49 to 75.89]

4. Secondary Outcome: Oxidative Stress Markers
Description: Change in F2-isoprostane levels
Time Frame: Change from baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Efavirenz | Rilpivirine
Number analyzed (Participants) | 14 | 12
pg/mL | 92.7 (178.6) | -101.4 (215.7)
Statistical Analysis 1: Comparison: Efavirenz vs Rilpivirine; Test type: Superiority or Other; p = 0.02, t-test, 2 sided; Mean Difference (Net) = -194.1, 95% CI 2-sided [-353.7 to -34.6]

ADVERSE EVENTS:
Time Frame: One month
Arm/Group | Efavirenz | Rilpivirine
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 17/20 | 11/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efavirenz (N=20) | Rilpivirine (N=20)
Dermatologic Abnormality (Skin and subcutaneous tissue disorders) | 2 | 2 — Rash or pruritis
CNS Abnormalities (Nervous system disorders) | 11 | 6 — Insomnia, Vivid Dreams, Drowsiness, Dizziness, Headache
Gastrointestinal Abnormalities (Gastrointestinal disorders) | 4 | 3 — Diarrhea, abdominal pain, nausea, vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No